CLINICAL TRIAL: NCT00661778
Title: An Open Label Study to Assess the Effect of First-line Treatment With Avastin in Combination With Docetaxel and Cisplatin on Progression-free Survival in Patients With Metastatic or Locally Advanced Non-small Cell Lung Cancer
Brief Title: A Study of Avastin (Bevacizumab) in Combination With Docetaxel and Cisplatin in Patients With Metastatic or Locally Advanced Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20081; 2006-005619-88 (EudraCT Number)
Record Dates: First submitted 2008-04-17; First posted 2008-04-18 (Estimated); Results first posted 2014-07-10 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Cisplatin; Docetaxel

ARMS (1):
- Bevacizumab + cisplatin + docetaxel (Experimental): Participants received bevacizumab 15 mg/kg intravenously (IV) followed by docetaxel 75 mg/kg IV in combination with cisplatin 75 mg/m^2 IV on Day 1 of each 3-week cycle for a maximum of 6 cycles. After completing the 6 cycles of combined chemotherapy, participants received bevacizumab 15 mg/kg IV until disease progression, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Bevacizumab; Drug: Cisplatin; Drug: Docetaxel

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab was supplied as a sterile liquid in glass vials.
  Other Names: Avastin
Drug: Cisplatin — Bevacizumab was supplied as a sterile liquid in glass vials.
Drug: Docetaxel — Bevacizumab was supplied as a sterile liquid in glass vials.
  Other Names: Taxotere

SUMMARY:
This study assessed the efficacy and safety of Avastin in combination with docetaxel and cisplatin as first-line treatment of patients with metastatic or locally advanced non-small cell lung cancer. Patients received Avastin 15 mg/kg intravenously (IV), docetaxel 75 mg/m^2, and cisplatin 75 mg/m^2 on Day 1 of each 3-week cycle for a maximum of 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, ≥ 18 years of age.
* Stage IIIb or IV non-small cell lung cancer.
* Chemotherapy-naive.

Exclusion Criteria:

* Previous treatment for non-small cell lung cancer.
* Previous malignant tumor within last 5 years, except for basal cell skin cancer or preinvasive cervical cancer.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to start of study.
* Recent or current chronic treatment with aspirin (> 325 mg/day).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- Spain (12):
  - Palma de Mallorca, Balearic Islands
  - Cadiz, Cadiz
  - Castellon, Castellon
  - Donostia / San Sebastian, Guipuzcoa
  - Alcalá de Henares, Madrid
  - Madrid, Madrid
  - Málaga, Malaga
  - Palencia, Palencia
  - Sagunto, Valencia
  - Valencia, Valencia
  - Valladolid, Valladolid
  - Zamora, Zamora

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The data listed in Participant Flow are for discontinuation from treatment, not discontinuation from the study. Data for discontinuation from the study are not available.
Period: Overall Study
Arm/Group | Bevacizumab + Cisplatin + Docetaxel
Started | 50
Completed | 0
Not Completed | 50
Not completed — Disease Progression | 23
Not completed — Adverse Event | 18
Not completed — Reason not Specified | 6
Not completed — Protocol Violation | 2
Not completed — Withdrawal of Consent | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: All enrolled participants who received at least 1 treatment.
Arm/Group | Bevacizumab + Cisplatin + Docetaxel
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.31 (9.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 38

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from enrollment in the study to the first documented disease progression using Response Evaluation Criteria In Solid Tumors (RECIST) or death from any cause, whichever occurred first.
Time Frame: Baseline to the end of the study (up to 4 years)
Population: Per protocol population: All participants who received at least 1 dose of study medication and had no major protocol deviations.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab + Cisplatin + Docetaxel
Number analyzed (Participants) | 49
Months | 8.95 [6.92 to 9.97]

2. Secondary Outcome: Percentage of Participants With an Objective Response
Description: An objective response was defined as a complete or partial response determined on 2 consecutive occasions ≥ 4 weeks apart using Response Evaluation Criteria in Solid Tumors (RECIST). Complete response was defined as the disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must be < 10 mm on the short axis. Partial response was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum.
Time Frame: Baseline to the end of the study (up to 4 years)
Population: Evaluable population: All participants who received at least 2 treatment cycles, have had all baseline lesions assessed on at least 1 occasion after receiving the 2nd treatment cycle, and have not had any major protocol violations.
Measure: Number; unit: Percentage of participants
Arm/Group | Bevacizumab + Cisplatin + Docetaxel
Number analyzed (Participants) | 46
Percentage of participants | 67.39

3. Secondary Outcome: Duration of the Objective Response
Description: Duration of the objective response is defined as the time from a complete or partial response to disease progression or death due to disease.
Time Frame: Baseline to the end of the study (up to 4 years)
Reporting Status: Not Posted

4. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from the first dose of study medication until death.
Time Frame: Baseline to the end of the study (up to 4 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Bevacizumab + Cisplatin + Docetaxel
Number analyzed (Participants) | 46
Months | 12.74 [9.48 to 17.79]

5. Secondary Outcome: 1-year Survival
Description: The probability of surviving 1 year was estimated using the Kaplan-Meier method.
Time Frame: Baseline to 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bevacizumab + Cisplatin + Docetaxel
Number analyzed (Participants) | 46
Percentage of participants | 53.46 [39.19 to 67.45]

ADVERSE EVENTS:
Description: Safety population: All enrolled participants who received at least 1 treatment and who satisfied all inclusion criteria and none of the exclusion criteria. One participant satisfied an exclusion criterion and was not included in the safety population.
Arm/Group | Bevacizumab + Cisplatin + Docetaxel
Serious Adverse Events (participants affected / at risk) | 26/49
Other Adverse Events (participants affected / at risk) | 48/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Cisplatin + Docetaxel (N=49)
Neutrophil count increased (Investigations) | 6
Positron emission tomography (Investigations) | 1
Decreased leukocyte count (Investigations) | 1
Respiratory tract infection (Infections and infestations) | 2
Oral candidiasis (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Wound evisceration (Injury, poisoning and procedural complications) | 1
Appendectomy (Surgical and medical procedures) | 1
Palpitations (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 3
Mucosal inflammation (General disorders) | 2
Reaction at the injection site (General disorders) | 1
Asthenia (General disorders) | 1
Death (General disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Cisplatin + Docetaxel (N=49)
Decreased hemoglobin (Investigations) | 21
High neutrophil count (Investigations) | 14
Decreased platelet count (Investigations) | 11
Elevated blood creatinine (Investigations) | 10
Decreased leukocyte count (Investigations) | 9
Gamma glutamyltransferase (Investigations) | 7
Elevated alanine aminotransferase (Investigations) | 4
Decreased total protein (Investigations) | 3
Decreased lymphocyte count (Investigations) | 3
Abnormal transaminases (Investigations) | 3
Elevated blood urea (Investigations) | 3
Urinary urobilin (Investigations) | 2
Decreased neutrophil count (Investigations) | 2
Elevated leukocyte count (Investigations) | 2
Increased blood alkaline phosphatase (Investigations) | 2
Elevated gamma glutamyl transferase (Investigations) | 2
Elevated blood lactate dehydrogenase (Investigations) | 2
Elevated blood bilirubin (Investigations) | 2
Blood urea (Investigations) | 1
Decreased monocyte count (Investigations) | 1
Hipofonesis (Investigations) | 1
Elevated triglycerides in blood (Investigations) | 1
Elevated ferritin in serum (Investigations) | 1
Positron emission tomography (Investigations) | 1
Alanine aminotransferase (Investigations) | 1
Abnormal coagulation test (Investigations) | 1
Increased international normalised ratio (Investigations) | 1
Prolonged activated partial thromboplastin time (Investigations) | 1
Decreased blood creatinine (Investigations) | 1
Decreased calcium in blood (Investigations) | 1
White blood count (Investigations) | 1
Lymphocyte count (Investigations) | 1
Elevated aspartate aminotransferase (Investigations) | 1
Respiratory tract infection (Infections and infestations) | 5
Infection (Infections and infestations) | 3
Respiratory tract infection (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Oral candidiasis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Parotiditis (Infections and infestations) | 1
Oral infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Anal abscess (Infections and infestations) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Wound evisceration (Injury, poisoning and procedural complications) | 1
Appendectomy (Surgical and medical procedures) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1
Palpitations (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 22
Onycholysis (Skin and subcutaneous tissue disorders) | 3
Ungueal toxicity (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Generalised erythema (Skin and subcutaneous tissue disorders) | 1
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 1
Cutaneous toxicity (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Hyperpigmentation of the skin (Skin and subcutaneous tissue disorders) | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Lymphopenia (Blood and lymphatic system disorders) | 2
Bone marrow depression (Blood and lymphatic system disorders) | 1
Amenorrhea (Reproductive system and breast disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 17
Hyperglycemia (Metabolism and nutrition disorders) | 11
Hyponatremia (Metabolism and nutrition disorders) | 7
Hypokalemia (Musculoskeletal and connective tissue disorders) | 5
Hypercholesterolemia (Metabolism and nutrition disorders) | 5
Hyperpotassemia (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Neuropathy (Nervous system disorders) | 13
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Decreased consciousness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 27
Nausea (Gastrointestinal disorders) | 19
Vomiting (Gastrointestinal disorders) | 18
Constipation (Gastrointestinal disorders) | 11
Dry mouth (Gastrointestinal disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 4
Odynophagia (Gastrointestinal disorders) | 2
Oesophagitis (Gastrointestinal disorders) | 2
Rectal bleeding (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Retching (Gastrointestinal disorders) | 1
Hematemesis (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 36
Mucosal inflammation (General disorders) | 21
Pyrexia (General disorders) | 15
Pain (General disorders) | 6
Asthenia (General disorders) | 3
Edema (General disorders) | 2
Reaction at the injection site (General disorders) | 2
Peripheral edema (General disorders) | 2
Chest pain (General disorders) | 2
Extravasation (General disorders) | 1
Death (General disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1
Pain in one extremity (Musculoskeletal and connective tissue disorders) | 1
Pain in the chest wall (Musculoskeletal and connective tissue disorders) | 1
Pain in sacrum (Musculoskeletal and connective tissue disorders) | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1
Increased lacrimation (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Anxiety (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 3
Disorientation (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 7
Hematuria (Renal and urinary disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 19
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Perforation of the nasal septum (Respiratory, thoracic and mediastinal disorders) | 1
Hiccupping (Respiratory, thoracic and mediastinal disorders) | 1
Orthopnea (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 8
Phlebitis (Vascular disorders) | 4
Deep vein thrombosis (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1
Flushing (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.